CLINICAL TRIAL: NCT04546932
Title: Lung-protective Mechanical Ventilation for Patients Undergoing Abdominal Laparoscopic Surgeries: A Randomized Controlled Trial
Brief Title: Lung-protective Mechanical Ventilation for Abdominal Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Collaborators: Vietnam National Cancer Hospital (Individual)
Responsible Party: Principal Investigator, Nguyen Trung Kien, Head of Center of Emergency, Critical Care Medicine and Clinical Toxicology, Military Hospital 103, Vietnam Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VMMU20193
Record Dates: First submitted 2020-08-20; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Mechanical Ventilation Complication
Keywords: Lung-protective mechanical ventilation; Low tidal volume; Positive end-expiratory pressure; Recruitment maneuvers

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to receive either lung-protective ventilation (LPV group) or conventional ventilation (CV group) at a ratio of 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An anesthesiologist who did not involve in the study set the ventilator in accordance with the protocol in the envelopes. Another anesthetist who was in charge of the patient collected data during surgery. The surgeons taking part in the procedures and patients were not informed of the ventilator setting. Physicians in post-anesthesia care unit who were not responsible for intraoperative care carried out the postoperative evaluation. The analysis of the postoperative chest X-ray was completed by a radiologist who was not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung-protective mechanical ventilation (Experimental): Vt=7 ml/kg IBW; an intraoperative 10 cmH2O in PEEP, recruitment maneuvers applying a stepwise increase in PEEP.
  Interventions: Procedure: Lung-protective mechanical ventilation
- Conventional mechanical ventilation (No Intervention): the tidal volume was set at 10 ml/kg IBW without PEEP and (recruitment maneuvers) RM

INTERVENTIONS:
Procedure: Lung-protective mechanical ventilation — Patients were provided with a tidal volume of 7 ml/kg IBW and an intraoperative 10 cmH2O in PEEP. Simultaneously, the alveoli were recruited applying a stepwise increase in PEEP (from 4 to 10 cmH2O for 3 breaths, 10 to 15 cmH2O for 3 breaths, and 15 to 20 cmH2O for 10 breaths) with maximum PIP = 50 cmH2O [24]. The recruitment maneuvers were performed right after intubation, 30 minutes after CO2 insufflation, then every hour, and finally before extubation.
  Arms: Lung-protective mechanical ventilation

SUMMARY:
This was a double-blind, randomized controlled clinical trial. 62 patients were randomly assigned to receive either lung-protective ventilation (LPV) with a tidal volume (Vt) of 7 ml/kg ideal body weight (IBW), 10 cmH2O positive end-expiratory pressure (PEEP) combined with regular recruitment maneuvers or conventional ventilation (CV) with a Vt of 10 ml/kg IBW, 0 cmH2O in PEEP and no recruitment maneuvers. The primary endpoints were the intraoperative fluctuation of Cdyn and Cstat, the intra- and postoperative changes in pulmonary oxygenation function including OI, A-aO2. The secondary endpoints were the alteration on chest x-ray, modified Clinical Pulmonary Infection Score (mCPIS), and the incidence of PPCs on the first postoperative day

DETAILED DESCRIPTION:
Study population. We performed a randomized, double-blind controlled trial at Vietnam National Cancer Hospital from January 2020 to July 2020. The trial protocol was approved by the medical ethics committee of Vietnam Military Medical University and Vietnam National Cancer Hospital, simultaneously written informed consent was obtained from all patients before inclusion.

Randomization and blinding technique. Participants were randomly assigned to receive either lung-protective ventilation (LPV group) or conventional ventilation (CV group) at a ratio of 1:1. The randomization was performed using the R program with the "runif", "as.integer", "int" and "replace" functions. As a result, a list of random numbers was created in each group. The patients were numbered according to their orders of hospital registration and then were allocated into the group of their numbers. The intervention protocol was stored in sealed, opaque numbered envelopes. An anesthesiologist who did not involve in the study set the ventilator in accordance with the protocol in the envelopes. Another anesthetist who was in charge of the patient collected data during surgery. The surgeons taking part in the procedures and patients were not informed of the ventilator setting. Physicians in post-anesthesia care unit who were not responsible for intraoperative care carried out the postoperative evaluation. The analysis of the postoperative chest X-ray was completed by a radiologist who was not involved in the study.

Standard procedure. All patients fasted for 12 hours before the procedure but still consumed clear water until 2 hours prior to surgery in order to avoid preoperative dehydration. Participants were premedicated with intravenous midazolam 1-2 mg 30 minutes before the surgery. In the operating room, a radical arterial cannula was inserted to monitor invasive blood pressure, collect blood gas sample, and measure the pulse pressure variation (PPV) index to guide intraoperative fluid therapy. The ASA standards for monitoring such as pulse oximeter, capnography, electrocardiography, thermometer were applied prior to the insertion of an epidural catheter at level T7-T12 for postoperative analgesia.

All patients received intravenous fentanyl 2 µg/kg, lidocaine 40 mg, propofol 2 mg/kg, and rocuronium 1 mg/kg for the induction. Intubation was performed 90 seconds after the administration of muscle relaxant and then 8 mg dexamethasone was injected. Anesthesia was maintained using sevoflurane of which the concentration was justified to achieve the end-tidal concentration within the range of 1,4-1,8 in oxygen and the PRST score less than 3. If the PRST score was greater than 3, then an additional bolus dose of 20-30 mg propofol and 25-50 µg fentanyl was injected along with increasing sevoflurane concentration. On the contrary, if signs of deep anesthesia were presented (PRST score=0, blood pressure decreased by more than 20% of the baseline values, bradycardia), then the sevoflurane concentration was cut down and 100 ml of crystalloid solution was rapidly infused within 2 minutes. A bolus dose of 100-200 µg phenylephrine was added if the blood pressure was still less than 20% of the baseline value in spite of these above-mentioned steps. Rocuronium was continuously infused at the rate of 10 µg/kg/min. The solution of bupivacaine 0,1% combined with fentanyl 2 µg/ml was infused via the epidural catheter at the rate of 5 ml/hour after a loading dose of 5 ml prior to skin incision. Normothermia was maintained during surgery. The pneumoperitoneum was implemented by CO2 insufflation at a pressure of 12 mmHg with room temperature in all patients. The intraoperative fluid was managed based on the goal-directed fluid therapy with a crystalloid solution. In brief, no additional fluids were provided if PPV was lower than 10%, otherwise, additional boluses of 250 ml ringer lactate solution were given over 10-15 minutes. After each bolus dose, PPV was re-assessed and further bolus was administered until reaching a PPV of lower than 10 %.

Intravenous 8 mg ondansetron was injected 30 minutes before the end of surgery to prevent postoperative nausea and vomiting. Rocuronium infusion was stopped 30 minutes before abdominal closure. The neuromuscular blockade was reversed in the postoperative care unit using intravenous neostigmine 40-60 µg/kg combined with atropine 0,5 mg. Patients were extubated when they met the extubation criteria (spontaneous tidal volume > 6 ml/kg and respiratory rate = 12-20 breath/minute, SpO2>95%, normocarbia, body temperature > 350C, positive gag reflexes and ability to follow a verbal command, hemodynamic stability without vasopressor support and ability to lift their heads and hold for 30 seconds [23]). Postoperative epidural analgesia for 48 hours was executed using bupivacaine 0,1% combined with fentanyl 2 µg/ml at a speed of infusion 5-10 ml/hour to maintain a visual analogue scale (VAS) score < 3. If the score was greater than 3, then a bolus dose 5 ml of the anesthetic solution was provided along with an increase in the speed of infusion. After extubation, patients were oxygenated via nasal cannula 3-5 ml/minute (1 ml/minute raises the FiO2 by 3%) to keep the SpO2>95%.

Ventilation protocol. Mechanical ventilation protocol was performed on the anesthesia machine GE healthcare carestation 620. The patient's ideal body weight was predefined according to formula: 45.5 + 0.91×[height(cm)-152.4] for women or 50 + 0.91×[height(cm)-152.4] for men. In both groups, the mechanical ventilation was set up at the volume-controlled mode, inspiration to expiration ratio of 1:2. After being lifted to 100% in the induction period, FiO2 was maintained at the level of 40% until extubation. Respiratory rate (starting with 18 breaths/minute) was justified to keep the end-tidal carbon dioxide (EtCO2) in the normal range of 35-40 mmHg. In the CV group, the tidal volume was set at 10 ml/kg IBW without PEEP and RM. In contrast, in the LPV group, patients were provided with a tidal volume of 7 ml/kg IBW and an intraoperative 10 cmH2O in PEEP. Simultaneously, in the LPV group, alveoli were recruited applying a stepwise increase in PEEP (from 4 to 10 cmH2O for 3 breaths, 10 to 15 cmH2O for 3 breaths, and 15 to 20 cmH2O for 10 breaths) with maximum PIP = 50 cmH2O [24]. The recruitment maneuvers were performed right after intubation, 30 minutes after CO2 insufflation, then every hour, and finally before extubation.

Data source and collection. The demographic characteristics including age, gender, height, weight, BMI, ASA physical status and history of coexisting diseases, and smoking were recorded. Vital signs (heart rate, blood pressure, SpO2, EtCO2, core temperature) were also recorded at 15 minutes intervals throughout the surgery. The volume of intravenous infusion (crystalloid, colloid solution), blood loss, urine output, total dose of anesthetics, fentanyl, and muscle relaxant were recorded as well. The dynamic compliance (Cdyn) was measured directly on the ventilator, while the static compliance (Cstat) was calculated in accordance with the pre-defined formula as Vt/(plateau pressure of the respiratory system - PEEP) with the plateau pressure measured during the normal ventilation setting using an inspiratory pause at 10% of the inspiratory time. Both types of pulmonary compliance were recorded at H0 (after intubation), H1 (30 minutes after pneumoperitoneum), H2 (1 hour after pneumoperitoneum), H3 (2 hours after pneumoperitoneum), Hkt (10 minutes after pneumoperitoneum stopped) and Hro (before extubation). Arterial blood samples were withdrawn from the radical arterial cannula for blood gas analysis before induction, 1 hour after pneumoperitoneum, and day 1 after operation. The pulmonary oxygenation index (OI) and the alveolar-arterial oxygen gradient (A-aO2) was calculated respectively as OI= PaO2/FiO2 and A-aO2= (PB-PH2O)×FiO2 -PaCO2/R - PaO2 where PB (atmospheric pressure) was 760 mmHg, PH2O (saturated vapor pressure at room temperature) was 47 mmHg, and the R (respiration quotient) was 0.8. SpO2 in the first postoperative day was measured in the room air (the nasal oxygen catheter was removed for 10 min) with the patient in bed. If SpO2 dropped to lower than 90%, the measurement was stopped and the supplemental oxygen was immediately re-provided via the nasal cannula.

Pre- and postoperative (day 1) chest radiography was obtained at the bedside and was analyzed in a blinded way by a radiologist who did not get involved in the study. Pathological chest X-ray was defined as the presence of at least one of the following: an increase in thickness of the interstitium, atelectasis, pleural effusion, localized or diffused infiltrates, and other chest radiological alterations.

Modified Clinical Pulmonary Infection Score (mCPIS). The modified original version of the Clinical Pulmonary Infection Score described by pelosi et al. (2008) was applied in the first postoperative day.

Incidence of postoperative pulmonary complications (PPCs). PPCs were defined by the European Perioperative Clinical Outcome (EPCO) definitions .

Primary and secondary endpoints. Our hypothesis was that the intraoperative lung-protective ventilation strategy could improve the pulmonary mechanics, oxygenation function, and ameliorate early postoperative pulmonary complications. The primary endpoints were the intraoperative fluctuation of Cdyn and Cstat, the intra- and postoperative changes in pulmonary oxygenation function including OI, A-aO2. The secondary endpoints were the alteration on chest x-ray, mCPIS, and the incidence of PPCs on the first postoperative day.

Statistical analysis. The sample size was calculated in accordance with the formula: n= (2×C)/δ2 +1 with δ=|µ1-µ2|/σ, where n is the sample size in each group, µ1= mean of OI in the LPV group, µ2 = mean of OI in the CV group, σ is the common standard deviation and c = 7.9 for 80% power. Based on the study of Xin Pi (2015) whose primary outcome was the OI after 2 hours of ventilation in the two groups was 382.21 ± 88.03 µg and 450.10 ± 70.29 µg respectively. Replacing µ1=382.21, µ2=450,10, σ=88,03 in the formula, n was equal to 27,5 for each group, which represented that the minimum sample size for each group was at least 28 patients.

Statistical analysis was completed using SPSS software version 20.0 (IBM, USA) on an intention-to-treat basis. Whether variables distributed normally was tested with the Kolmogorov-Smirnov and Shapiro-Wilk test. Continuous variables were compared applying either Student's t-test or the Mann-Whitney U test, depending on the characteristics of the distribution of the variable, and consequently were presented as mean ± SD or median and interquartile range (25-75%) as appropriate. As for categorical variables, the χ2 test was employed for comparison and the Fisher exact test was used for small frequencies. All the tests were two-tailed, and statistical significance was accepted at p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal laparoscopic surgeries under general anesthesia with an expected duration of greater than 2 hours.
* Age more than 18 years.
* American Society of Anesthesiologists (ASA) physical status I-III.
* A body mass index (BMI) less than 30 kg/m2.

Exclusion Criteria:

* Individuals who refused to participate in the study.
* Patients with preexisting cardiac or pulmonary comorbidities (for instance heart failure, intractable shock, chronic obstructive pulmonary disease, asthma, pulmonary infection, bronchiectasis, pulmonary metastases ).
* Any preexisting abnormalities on chest X-ray or spirometry.
* Neuromuscular disease.
* Liver cirrhosis (Child B or C).
* Chronic renal failure with dialysis.
* A need for prolonged mechanical ventilation after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Changes in intraoperative pulmonary dynamic compliance | H0 (after intubation), H1 (30 minutes after pneumoperitoneum), H2 (1 hour after pneumoperitoneum), H3 (2 hours after pneumoperitoneum), Hkt (10 minutes after pneumoperitoneum stopped) and Hro (before extubation)
  At a specific time point, the dynamic compliance (Cdyn in ml/cmH2O) was measured directly on the ventilator. Changes in Cdyn were recorded at H0 (after intubation), H1 (30 minutes after pneumoperitoneum), H2 (1 hour after pneumoperitoneum), H3 (2 hours after pneumoperitoneum), Hkt (10 minutes after pneumoperitoneum stopped) and Hro (before extubation).
Changes in intraoperative pulmonary static compliance | H0 (after intubation), H1 (30 minutes after pneumoperitoneum), H2 (1 hour after pneumoperitoneum), H3 (2 hours after pneumoperitoneum), Hkt (10 minutes after pneumoperitoneum stopped) and Hro (before extubation)
  At a specific time point, the static compliance (Cstat in ml/cmH2O)) was calculated in accordance with the pre-defined formula as Vt (ml)/[plateau pressure of the respiratory system (cmH2O) - PEEP(cmH2O)] with the plateau pressure was measured during the normal ventilation setting using an inspiratory pause at 10% of the inspiratory time. Changes in Cstat were recorded at H0 (after intubation), H1 (30 minutes after pneumoperitoneum), H2 (1 hour after pneumoperitoneum), H3 (2 hours after pneumoperitoneum), Hkt (10 minutes after pneumoperitoneum stopped) and Hro (before extubation)
Changes in pre-, intra- and postoperative oxygenation index (OI) | before induction, 1 hour after pneumoperitoneum, and day 1 after operation
  At a specific time point, the pulmonary oxygenation index (OI in mmHg) was calculated by the pre-defined formula: OI (mmHg) = PaO2 (mmHg)/FiO2 (%) where PaO2 was partial pressure of oxygen in arterial blood obtained by blood gas analysis and FiO2 was fraction of inspired oxygen.
  Changes in OI were recorded before induction, 1 hour after pneumoperitoneum, and day 1 after operation.
Changes in pre-, intra- and postoperative alveolar-arterial oxygen gradient (A-aO2) | before induction, 1 hour after pneumoperitoneum, and day 1 after operation
  At a specific time point, the alveolar-arterial oxygen gradient (A-aO2 in mmHg) was calculated as A-aO2 (mmHg) = (PB-PH2O)×FiO2 -PaCO2/R - PaO2 where PB (atmospheric pressure) was 760 mmHg, PH2O (saturated vapor pressure at room temperature) was 47 mmHg, and the R (respiration quotient) was 0.8, PaCO2 in mmHg and PaO2 in mmHg.
  Changes in A-aO2 were recorded.before induction, 1 hour after pneumoperitoneum, and day 1 after operation.

SECONDARY OUTCOMES:
Chest radiography on day 1 after surgery | day 1 after surgery
  Postoperative (day 1) chest radiography was obtained at the bedside and was analyzed by a radiologist who did not get involved in the study. Pathological chest X-ray was defined as the presence of at least one of the followings: an increase in thickness of the interstitium, atelectasis, pleural effusion, localized or diffused infiltrates.
Modified Clinical Pulmonary Infection Score (mCPIS) | day 1 after surgery
  Modified Clinical Pulmonary Infection Score (mCPIS) was calculated for each patient on the first day after surgery. The modified original version of the Clinical Pulmonary Infection Score was described by pelosi et al. (2008) measuring based on body temperature, blood leukocytes, tracheal secretions, the ratio of PaO2/FiO2 and chest radiograph
Incidence of postoperative pulmonary complications (PPCs) | day 1 after surgery
  Incidence of postoperative pulmonary complications (PPCs in percentage) was measured in each group. PPCs were defined by the European Perioperative Clinical Outcome (EPCO) definitions including respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis.

CONTACTS AND LOCATIONS:
Overall Officials: Kien T Nguyen, PhD, Principal Investigator — Critical Care Medicine and ClinicalToxicology, Military Hospital 103
Locations (1):
- Department of Anesthesia and Pain Medicine, Vietnam National Cancer Hospital, Hanoi, Ha Dong District, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD will be shared to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: no criteria

REFERENCES:
- [Result] Pi X, Cui Y, Wang C, Guo L, Sun B, Shi J, Lin Z, Zhao N, Wang W, Fu S, Li E. Low tidal volume with PEEP and recruitment expedite the recovery of pulmonary function. Int J Clin Exp Pathol. 2015 Nov 1;8(11):14305-14. eCollection 2015. PMID 26823746
- [Result] Severgnini P, Selmo G, Lanza C, Chiesa A, Frigerio A, Bacuzzi A, Dionigi G, Novario R, Gregoretti C, de Abreu MG, Schultz MJ, Jaber S, Futier E, Chiaranda M, Pelosi P. Protective mechanical ventilation during general anesthesia for open abdominal surgery improves postoperative pulmonary function. Anesthesiology. 2013 Jun;118(6):1307-21. doi: 10.1097/ALN.0b013e31829102de. PMID 23542800
- [Result] Liu J, Meng Z, Lv R, Zhang Y, Wang G, Xie J. Effect of intraoperative lung-protective mechanical ventilation on pulmonary oxygenation function and postoperative pulmonary complications after laparoscopic radical gastrectomy. Braz J Med Biol Res. 2019;52(6):e8523. doi: 10.1590/1414-431x20198523. Epub 2019 Jun 3. PMID 31166383
- [Result] Sprung J, Whalen FX, Comfere T, Bosnjak ZJ, Bajzer Z, Gajic O, Sarr MG, Schroeder DR, Liedl LM, Offord CP, Warner DO. Alveolar recruitment and arterial desflurane concentration during bariatric surgery. Anesth Analg. 2009 Jan;108(1):120-7. doi: 10.1213/ane.0b013e31818db6c7. PMID 19095839
- [Result] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Result] Futier E, Constantin JM, Petit A, Jung B, Kwiatkowski F, Duclos M, Jaber S, Bazin JE. Positive end-expiratory pressure improves end-expiratory lung volume but not oxygenation after induction of anaesthesia. Eur J Anaesthesiol. 2010 Jun;27(6):508-13. doi: 10.1097/EJA.0b013e3283398806. PMID 20404729
- [Result] Hazebroek EJ, Haitsma JJ, Lachmann B, Bonjer HJ. Mechanical ventilation with positive end-expiratory pressure preserves arterial oxygenation during prolonged pneumoperitoneum. Surg Endosc. 2002 Apr;16(4):685-9. doi: 10.1007/s00464-001-8174-y. Epub 2001 Dec 31. PMID 11972215
- [Result] Whalen FX, Gajic O, Thompson GB, Kendrick ML, Que FL, Williams BA, Joyner MJ, Hubmayr RD, Warner DO, Sprung J. The effects of the alveolar recruitment maneuver and positive end-expiratory pressure on arterial oxygenation during laparoscopic bariatric surgery. Anesth Analg. 2006 Jan;102(1):298-305. doi: 10.1213/01.ane.0000183655.57275.7a. PMID 16368847
- [Result] Haliloglu M, Bilgili B, Ozdemir M, Umuroglu T, Bakan N. Low Tidal Volume Positive End-Expiratory Pressure versus High Tidal Volume Zero-Positive End-Expiratory Pressure and Postoperative Pulmonary Functions in Robot-Assisted Laparoscopic Radical Prostatectomy. Med Princ Pract. 2017;26(6):573-578. doi: 10.1159/000484693. Epub 2017 Oct 31. PMID 29131002
- [Result] Pelosi P, Barassi A, Severgnini P, Gomiero B, Finazzi S, Merlini G, d'Eril GM, Chiaranda M, Niederman MS. Prognostic role of clinical and laboratory criteria to identify early ventilator-associated pneumonia in brain injury. Chest. 2008 Jul;134(1):101-8. doi: 10.1378/chest.07-2546. Epub 2008 Apr 10. PMID 18403669
- [Derived] Nguyen TK, Nguyen VL, Nguyen TG, Mai DH, Nguyen NQ, Vu TA, Le AN, Nguyen QH, Nguyen CT, Nguyen DT. Lung-protective mechanical ventilation for patients undergoing abdominal laparoscopic surgeries: a randomized controlled trial. BMC Anesthesiol. 2021 Mar 30;21(1):95. doi: 10.1186/s12871-021-01318-5. PMID 33784987